CLINICAL TRIAL: NCT04206761
Title: Xenon MRI Probing vEntilation Response to Triple Therapy (QVM149)
Brief Title: Investigating the Effects of QVM149 on MRI Ventilation Defects
Acronym: XPERTT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: issues related to Covid-19 restrictions/shutdowns
Sponsor: Dr. Grace Parraga (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Dr. Grace Parraga, Professor, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROB0045
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2020-10

CONDITIONS: Asthma
Keywords: QVM149; Indacaterol; Glycopyrronium; Mometasone; Xenon; Triple Therapy
MeSH Terms: conditions — Asthma | interventions — indacaterol

STUDY DESIGN:
Intervention Model Description: A single site, two arm, randomized, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment - QVM149 (Experimental): Participants will complete a two week treatment with QVM149 (indacaterol acetate/glycopyrronium bromide/mometasone furoate) 150/50/160 μg delivered as powder in hard capsules via Breezhaler, a breath-activated device which will deliver a specific dose of medication via inhalation.
  Interventions: Drug: QVM149
- Control (Active Comparator): Participants will continue their clinically prescribed treatment with a high dose dual therapy of Inhaled Corticosteroid (ICS)/Long-Acting Beta2-Agonist (LABA) in any approved drug formulation and delivery device for the treatment period of two weeks. (Participants will continue receiving high dose ICS/LABA therapy at the same dose and in the same formulation as at baseline).
  Interventions: Drug: High Dose Dual Therapy (ICS/LABA)

INTERVENTIONS:
Drug: QVM149 — QVM149 is an investigational drug consisting of 150μg indacaterol acetate, 50μg glycopyrronium bromide and 160μg mometasone furoate. The drug is delivered as powder in hard capsules via Breezhaler, a breath-activated device which will deliver a specific dose of medication
  Other Names: indacaterol acetate/glycopyrronium bromide/mometasone furoate
  Arms: Treatment - QVM149
Drug: High Dose Dual Therapy (ICS/LABA) — High dose inhaled corticosteroid (ICS)/long-acting beta2-agonist (LABA) in any approved drug formulation and delivery device.
  Arms: Control

SUMMARY:
The purpose of this study is to compare treatment with QVM149, an inhaler that contains three types of asthma medications compared to an inhaler that contains two types of asthma medications. Both inhalers contain an inhaled corticosteroid, which reduces inflammation in the lungs, and a medication that helps to open up the airways. The investigational inhaler, QVM149, contains a third medication that also works to open up the airways. The investigators will measure the difference in these two treatments with magnetic resonance imaging (MRI) using a special technique using xenon gas to show how gas spreads in the lungs. In healthy lungs, the gas fills the lungs evenly, but in unhealthy lungs, the gas may fill the lungs unevenly and they will appear patchy. The patchy areas are called ventilation defects. A CT of the chest will be done to assess the structure of the lungs. The investigators will also use lung function testing and questionnaires to evaluate the differences between these therapies.

DETAILED DESCRIPTION:
A single site, two arm, randomized, open-label study in participants with asthma, who demonstrate visually obvious ventilation defects despite being on ICS/LABA was chosen to evaluate the capability of QVM149 150/50/160 μg once daily as compared to high dose dual therapy (ICS/LABA) to improve ventilation heterogeneity. According to the design of the study, hyperpolarized Xenon-129 (129Xe) will be used to measure ventilation defects in asthma participants as ventilation defect percent (VDP). A low-dose chest CT acquired within a few minutes of MRI will provide a way to measure both airway and parenchymal abnormalities. The selection of the QVM149 150/50/160 μg was made in order to keep the ICS dose equipotent to baseline therapy and to the active comparator arm and to directly compare the addition of a long-acting muscarinic antagonist (LAMA) versus continuing the therapy with high dose dual therapy (ICS/LABA).

This study will be a single site, two arm, randomized, open-label study with the following treatment:

* Treatment A: 2-week treatment with Indacaterol/Glycopyrronium/Mometasone 150/50/160 μg delivered as powder in hard capsules via Breezhaler, a breath-activated device which will deliver a specific dose of medication.
* Treatment B: 2-week treatment with high dose dual therapy (ICS/LABA) in any approved drug formulation and delivery device. (Continue receiving high dose ICS/LABA therapy at the same dose and in the same formulation as at baseline).

The study will consist of a screening/inclusion period of 1-5 days, followed by a treatment period of 14 days. The evaluation team including MRI observers will be blinded to treatment.

At Visit 101, informed consent will be obtained before any study related assessments or procedures are performed. Asthma medications and eligibility criteria will be reviewed. Furthermore, at Visit 101, safety assessments including electrocardiography (ECG), hematology, blood chemistry, urinalysis, and spirometry to test reversibility will be performed. Once the above criteria are met, participants will move on to Visit 102.

At Visit 102 all additional assessments, including MRI to detect visually obvious ventilation defects, low-dose chest CT, and Pulmonary Function Test assessments including spirometry, plethysmography, Lung Clearance Index (LCI) and Forced Oscillation Technique (FOT) will be conducted. Participants who qualify will then be randomized and entered into the 14 days treatment period and continue with the assessments according to study protocol. Participants will be supplied with open-label Indacaterol/Glycopyrronium/ Mometasone 150/50/160 μg o.d. delivered as powder in hard capsules via Breezhaler or continue with their previously prescribed high dose dual therapy (ICS/LABA) in any approved drug formulation and delivery device, which will be used during the study treatment period and stopped at Visit 201.

Upon completion of the study treatment period at Visit 201, all participants will undergo post-treatment assessments, including MRI, pre- and post-salbutamol pulmonary function testing including spirometry, plethysmography, LCI, FOT, and asthma questionnaires.

A final visit, Visit 301 will be scheduled for safety assessments. All participants will undergo vital signs, spirometry, ECG, bloodwork and urinalysis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be directly obtained from legally competent participants before any study- related assessment is performed.
* Male and female adult participant ≥ 18 years of age and ≤ 80 years of age.
* Participants with a confirmed clinical diagnosis of asthma by a respirologist for a period of at least 6 months prior to Visit 101.
* Participants who demonstrate reversibility in FEV1 by one of :

  1. Increase in forced expiratory volume in one second (FEV1) of ≥ 12% and 200 ml 15 to 30 minutes after administration of 400μg salbutamol at Visit 101
  2. Documented increase in FEV1 of ≥ 12% and 200 ml 15 to 30 minutes after administration of 400μg salbutamol in past 24 months
  3. Documented increase in FEV1 of ≥ 12% and 200 ml after treatment for asthma (e.g. treatment with ICS) in past 24 months
  4. Documented positive methacholine challenge in past 24 months
* Participants who have used high dose dual therapy (ICS/LABA) for asthma for at least 3 months and at a stable dose equivalent to high dose ICS for at least 1 month prior to Visit 101 (please refer to Table 1-1 for ICS dosages).
* Participants with visually obvious MRI ventilation defects at Visit 102.
* Pre-bronchodilator FEV1 of < 85% of the predicted normal value for the participant after withholding bronchodilators prior to spirometry at Visit 101.

Exclusion Criteria:

* Participants meeting contraindications for undergoing an MRI such as participants with MRI-sensitive implants, tattoos with MRI-sensitive dye and severe claustrophobia.
* Currently smoking or vaping any substance (e.g. nicotine, cannabis) at Visit 101 or within 12 months of visit 101.
* Ex-smoker of nicotine or cannabis with a smoking history of ≥ 10 pack years or 20 joint years (Note: 1 pack is equivalent to 20 cigarettes. 10 pack years = 1 pack /day x 10 yrs., or ½ pack/day x 20 yrs. 1 joint year is equivalent to 1 joint/day x 1 year)
* Participants diagnosed with Chronic Obstructive Pulmonary Disease (COPD). Diagnoses of asthma- COPD overlap syndrome may be eligible.
* Participants who have had an asthma attack/exacerbation requiring systemic steroids, hospitalization and/or emergency room visit within 6 weeks of Visit 101 or a respiratory tract infection requiring antibiotics within 4 weeks prior to Visit 101. If participants experience an asthma attack/exacerbation requiring systemic steroids or hospitalization or emergency room visit between Visit 101 and Visit 201, they will be withdrawn from the study but may be re-screened 4 weeks after recovery from the exacerbation.
* Participants treated with a LAMA for asthma within 3 months prior to Visit 101.
* Participants with narrow-angle glaucoma, symptomatic benign prostatic hyperplasia (BPH) or bladder- neck obstruction or severe renal impairment or urinary retention. BPH participants who are stable on treatment can be considered.
* Participants with a history of chronic lung diseases other than asthma, including (but not limited to) sarcoidosis, interstitial lung disease, cystic fibrosis, clinically significant bronchiectasis and active tuberculosis.
* Use of other investigational drugs within 30 days (e.g. small molecules) / or until the expected pharmacodynamic effect has returned to baseline (e.g. biologics), whichever is longer.
* History of hypersensitivity to any of the study treatments or its excipients or to other drugs of similar chemical classes.
* Participants with paroxysmal (e.g., intermittent) atrial fibrillation are excluded. Participants with persistent atrial fibrillation as defined by continuous atrial fibrillation for at least 6 months and controlled with a rate control strategy (i.e., selective beta blockers, calcium channel blocker, digoxin or ablation therapy) for at least 6 months may be considered for inclusion. In such participants, atrial fibrillation must be present at Visit 101 with a resting ventricular rate < 100/min.
* Participants with a history of myocardial infarction within 12 months prior to Visit 101.
* Concomitant use of agents known to prolong the QT interval unless it can be discontinued for the duration of study. Decisions about the discontinuation of such agents will be made between the Qualified Investigator and participant.
* Participants with a history of long QT syndrome or whose QTc measured at Visit 101 (Fridericia method) is prolonged (> 450 msec for males and > 460 msec for females). These participants may not be rescreened.
* Participants with a history of lactose intolerance and hypersensitivity to any of the study drugs or its excipients, or to similar drugs within the class including untoward reactions to sympathomimetic amines or inhaled medication or any component thereof.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of study treatment and follow-up period. Highly effective contraception methods include:

  1. True sexual abstinence with male partner(s) (when this is in line with the preferred and usual lifestyle of the participant). Periodic abstinence (e.g., calendar, ovulation, symptom-thermal, post ovulation methods) and withdrawal are not acceptable methods of contraception.
  2. Female sterilization (have had surgical tubal ligation, bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  3. Vasectomized male partner(s) (at least 6 months prior to Visit 101).
  4. Use hormonal contraception with failure rate <1% (e.g. oral contraceptive pill, Depo-Provera™ injections, Erva Patch™ or Nuvaring™).
  5. Placement of an MRI safe intrauterine device (IUD) or intrauterine system (IUS).

In case of use of hormonal contraception, women should have been stable on the same pharmacological agent for a minimum of 3 months before Visit 101. Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of childbearing potential.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline airway function measured using 129-Xenon MRI ventilation defect percent at the end of 2 weeks of treatment with QVM149 150/50/160 μg once daily | Day 0 and 14
  Change in VDP
Difference in change from baseline airway function measured using 129-Xenon MRI ventilation defect percent after 2 weeks use of QVM149 150/50/160 μg once daily compared to high dose dual therapy (ICS/LABA) | Day 0 and 14
  Difference in change in VDP

SECONDARY OUTCOMES:
Explore univariate correlation and linear regression of MRI ventilation defect percent and forced expiration volume in one second. | Day 14
  The relationship between ventilation defect percent and forced expiration volume in one second will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary function and structure.
Explore univariate correlation and linear regression of MRI ventilation defect percent and forced vital capacity | Day 14
  The relationship between ventilation defect percent and forced vital capacity will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary function and structure.
Explore univariate correlation and linear regression of MRI ventilation defect percent and lung volumes | Day 14
  The relationship between ventilation defect percent and lung volumes will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary function and structure.
Explore univariate correlation and linear regression of MRI ventilation defect percent and forced oscillation technique | Day 14
  The relationship between ventilation defect percent and forced oscillation technique will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary function, structure and inflammation.
Explore univariate correlation and linear regression of MRI ventilation defect percent and lung clearance index | Day 14
  The relationship between ventilation defect percent and lung clearance index will be assessed using univariate correlation analysis and linear regression. This information gives insight into the relationship between pulmonary function and structure.
Explore univariate correlation and linear regression of MRI ventilation defect percent and asthma control as measured by the Asthma Control Questionnaire | Day 14
  The relationship between ventilation defect percent and asthma control, as measured by the Asthma Control Questionnaire (ACQ-6) will be assessed using a univariate correlation analysis and linear regression. The ACQ-6 is scored from 0 to 6, with higher scores indicating more uncontrolled asthma.
Explore univariate correlation and linear regression of MRI ventilation defect percent and asthma-related quality of life as measured by the Asthma Quality of Life Questionnaire | Day 14
  The relationship between ventilation defect percent and asthma-related quality of life as measured by the Asthma Quality of Life Questionnaire with Standardised Activities (AQLQ(S)) will be assessed using a univariate correlation analysis and linear regression. The AQLQ(S) is scored from 1-7, with lower scores indicating more severe impairment.
Explore univariate correlation and linear regression of MRI ventilation defect percent and daily life and perceived well-being as measured by the St. George's Respiratory Questionnaire | Day 14
  The relationship between ventilation defect percent and daily life and perceived well-being as measured by the St. George's Respiratory Questionnaire (SGRQ) will be assessed using univariate correlation analysis and linear regression. The SGRQ is scored from 0-100 with higher scores indicating more limitations.
Change from baseline forced expiration volume in one second | Day 0 and 14
  Indicator of pulmonary function
Difference in change from baseline forced expiration volume in one second after use of QVM149 compared to high dose dual therapy. | Day 0 and 14
  Indicator of pulmonary function
Change from baseline forced vital capacity | Day 0 and 14
  Indicator of pulmonary function
Difference in change from baseline forced vital capacity after use of QVM149 compared to high dose dual therapy. | Day 0 and 14
  Indicator of pulmonary function
Change from baseline residual volume. | Day 0 and 14
  Indicator of pulmonary function
Difference in change from baseline residual volume after use of QVM149 compared to high dose dual therapy. | Day 0 and 14
  Indicator of pulmonary function
Change from baseline total lung capacity. | Day 0 and 14
  Indicator of pulmonary function
Difference in change from baseline total lung capacity after use of QVM149 compared to high dose dual therapy. | Day 0 and 14
  Indicator of pulmonary function
Change from baseline forced oscillation technique | Day 0 and 14
  Indicator of pulmonary function and inflammation
Difference in change from baseline forced oscillation technique after use of QVM149 compared to high dose dual therapy. | Day 0 and 14
  Indicator of pulmonary function and inflammation
Change from baseline lung clearance index | Day 0 and 14
  Indicator of pulmonary function
Difference in change from baseline lung clearance index after use of QVM149 compared to high dose dual therapy. | Day 0 and 14
  Indicator of pulmonary function
Change from baseline in asthma control | Day 0 and 14
  Asthma Control Questionnaire (ACQ-6) is used to evaluate asthma control. The ACQ-6 is scored from 0 to 6, with higher scores indicating more severely uncontrolled asthma.
Difference in change from baseline in asthma control after use of QVM149 compared to high dose dual therapy. | Day 0 and 14
  Asthma Control Questionnaire (ACQ-6) is used to evaluate asthma control. The ACQ-6 is scored from 0 to 6, with higher scores indicating more severely uncontrolled asthma.
Change from baseline in asthma-related quality of life | Day 0 and 14
  Asthma Quality of Life Questionnaire with Standardised Activities (AQLQ(S)) evaluates asthma-related quality of life. The AQLQ(S) is scored from 1-7, with lower scores indicating more severe impairment.
Difference in change from baseline in asthma-related quality of life after use of QVM149 compared to high dose dual therapy. | Day 0 and 14
  Asthma Quality of Life Questionnaire with Standardised Activities (AQLQ(S)) evaluates asthma-related quality of life. The AQLQ(S) is scored from 1-7, with lower scores indicating more severe impairment.
Change from baseline in daily life and perceived well-being as measured by the St. George's Respiratory Questionnaire | Day 0 and 14
  Asthma Quality of Life Questionnaire with Standardised Activities (AQLQ(S)) evaluates asthma-related quality of life. The AQLQ(S) is scored from 1-7, with lower scores indicating more severe impairment.
Difference in change from baseline in daily life and perceived well-being as measured by the St. George's Respiratory Questionnaire after use of QVM149 compared to high dose dual therapy. | Day 0 and 14
  Asthma Quality of Life Questionnaire with Standardised Activities (AQLQ(S)) evaluates asthma-related quality of life. The AQLQ(S) is scored from 1-7, with lower scores indicating more severe impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario
Locations (1):
- Robarts Research Insitute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No